CLINICAL TRIAL: NCT02198040
Title: Physiotherapy in the Treatment of Elbow Hemophilic Arthropathy: Manual Therapy vs Educational Physiotherapy. A Pilot Sudy
Brief Title: Physiotherapy in the Haemophilic Arthropathy of the Elbow.
Acronym: ELBOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELBOW; ELBOW
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2016-12

CONDITIONS: Patients With Hemophilia
Keywords: Elbow; Joint disease; Hemophilia; Physiotherapy modalities
MeSH Terms: conditions — Joint Diseases; Hemophilia A | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual Therapy group (Experimental): The treatment of this group consisted of two sessions per week, one hour each. We used joint traction, passive muscles stretching and Proprioceptive Neuromuscular Facilitation
  Interventions: Other: Manual Therapy
- Educational group (Experimental): The treatment had education and home daily exercises for the improvement of the range of motion, biceps strength, perimeter of arm and the perception of pain in patients with haemophilia and arthropathy of the elbow.
  Interventions: Other: Educational group
- Control group (No Intervention): The control group did not receive any intervention. The patients in this group were assessed by the same reviewers (blinded to the study conditions) and under the same conditions, that patients in the experimental groups.

INTERVENTIONS:
Other: Manual Therapy — * 5 minutes. Termotherapy shalow to 50 cm away from the elbow, using a bulb of 250w.
  * 15 minutes. Joint traction of elbow, in submaximal mobility amplitude with distal fixation of humerus and proximal fixation of radius and ulna in neutral position of forearm. Joint traction in I-II degree of flexion and extension submaximal of elbow.
  * 15 minutes. Passive muscle stretching (within the limits of mobility).
  * 15 minutes. Proprioceptive neuromuscular facilitation (PNF) of upper limb, from the abduction, flexion and external rotation of shoulder.
  * 10 minutes. Local cryotherapy with ice bag and protection between it and the skin
  Arms: Manual Therapy group
Other: Educational group — * Theory: Introduction to hemophilia: clinic and treatment; Anatomy and biomechanics of elbow; Anatomy of elbow musculature. Function of muscles and haematomas treatment; Haemarthrosis, synovitis and arthropathy: clinical manifestations and treatment; Proprioception: definition and importance in hemophilia; and Physical activity and sport: risks and benefits.
  * Practice: exercises in favor of gravity; isometric and isotonic exercises of elbow; active exercises for mobility and pain management; elbow proprioception exercises; and swimming technique.
  Arms: Educational group

SUMMARY:
The aim of this study is to assess the effectiveness of two treatments of Physiotherapy: one with joint traction, passive muscles stretching and Proprioceptive Neuromuscular Facilitation (PNF), and the other with education sessions and home exercises, for the improvement of the ROM, biceps strength, perimeter of arm and the perception of pain in PwH and arthropathy of the elbow.

DETAILED DESCRIPTION:
The intervention was carried out during twelve weeks, performing evaluations before and after treatment, and six months of finalizing this. The treatment of MT group consisted of two sessions per week, one hour each, and the treatment of group E consisted in a session for 90 minutes every two weeks, with daily home exercises. The control group (group C) did not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients diagnosed with hemophilia A or B
* Patients with hemophilic arthropathy in one or both elbows

Exclusion Criteria:

* Patients with another medical diagnosis (eg, Von Willebrand's disease)
* Patients with presence of antibodies to FVIII or FIX (inhibitors)
* Patients who had a haemarthrosis of elbow during the study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RUBEN CUESTA-BARRIUSO, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad de Murcia, Murcia, Spain

REFERENCES:
- [Derived] Cuesta-Barriuso R, Gomez-Conesa A, Lopez-Pina JA. Manual and educational therapy in the treatment of hemophilic arthropathy of the elbow: a randomized pilot study. Orphanet J Rare Dis. 2018 Sep 3;13(1):151. doi: 10.1186/s13023-018-0884-5. PMID 30176883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 patients Hemophilia of the Association of Murcia were recruited between January to October 2013
Pre-assignment Details: 28 patients who met the exclusion criteria. Only one declined to participate for personal reasons.
Groups:
- Manual Therapy Group: The treatment of this group consisted of two sessions per week, one hour each. Manual Therapy: - 5 minutes. Termotherapy shalow to 50 cm away from the elbow, using a bulb of 250w.
  * 15 minutes. Joint traction of elbow, in submaximal mobility amplitude with distal fixation of humerus and proximal fixation of radius and ulna in neutral position of forearm. Joint traction in I-II degree of flexion and extension submaximal of elbow.
  * 15 minutes. Passive muscle stretching (within the limits of mobility). Compression technique, passive muscle stretching and relaxation in biceps and triceps.
  * 15 minutes. Proprioceptive neuromuscular facilitation (PNF) of upper limb, from the abduction, flexion and external rotation of shoulder with extension of elbow and dorsal flexion of wrist, to adduction, internal rotation of shoulder with flexion of elbow and palmar flexion of wrist and fingers.
  * 10
- Educational Gruop: The treatment had education and home daily exercises for the improvement of the range of motion, biceps strength, perimeter of arm and the perception of pain in patients with haemophilia and arthropathy of the elbow.
  Educational group: - Theory: Introduction to hemophilia: clinic and treatment; Anatomy and biomechanics of elbow; Anatomy of elbow musculature. Function of muscles and haematomas treatment; Haemarthrosis, synovitis and arthropathy: clinical manifestations and treatment; Proprioception: definition and importance in hemophilia; and Physical activity and sport: risks and benefits.
  - Practice: exercises in favor of gravity; isometric and isotonic exercises of elbow; active exercises for mobility and pain management; elbow proprioception exercises; and swimming technique.
Period: Overall Study
Arm/Group | Manual Therapy Group | Educational Gruop | Control Group
Started | 9 | 9 | 9
Completed | 9 | 8 | 8
Not Completed | 0 | 1 | 1
Not completed — Work reasons | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Manual Therapy Group: The treatment of this group consisted of two sessions per week, one hour each.
  Manual Therapy: - 5 minutes. Termotherapy shalow to 50 cm away from the elbow, using a bulb of 250w.
  * 15 minutes. Joint traction of elbow, in submaximal mobility amplitude with distal fixation of humerus and proximal fixation of radius and ulna in neutral position of forearm. Joint traction in I-II degree of flexion and extension submaximal of elbow.
  * 15 minutes. Passive muscle stretching (within the limits of mobility). Compression technique, passive muscle stretching and relaxation in biceps and triceps.
  * 15 minutes. Proprioceptive neuromuscular facilitation (PNF) of upper limb, from the abduction, flexion and external rotation of shoulder with extension of elbow and dorsal flexion of wrist, to adduction, internal rotation of shoulder with flexion of elbow and palmar flexion of wrist and fingers.
  * 10 minutes. Local cryotherapy with ice bag and protection between it and the skin
- Total: Total of all reporting groups
Arm/Group | Manual Therapy Group | Educational Gruop | Control Group | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 27
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 9 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Spain | 9 | 9 | 9 | 27
Radiological joint deterioration [Mean (Standard Deviation); unit: units on a scale] — Radiological joint deterioration of elbows with Pettersson score. Mean score (and standard deviation) for elbow joint evaluated in patients enrolled in the study. This scale has a range from 0 to 13 points (0 indicates no joint damage and 13 indicates maximum joint damage) to assess the hemophilic arthropathy.
  units on a scale | 9.63 (1.62) | 8.50 (3.40) | 7.57 (2.90) | 8.61 (2.809)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Range of Motion of Elbow
Description: Measurement the changes of flexion and extension of elbow (in degrees) using a universal goniometer. We were taken as anatomical references, those specified by Querol et al, using the zero-method-reference for the mobile arm goniometer as indicated Norkin et al.
Time Frame: Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
Population: It has made an analysis by intention to treat with the 27 patients included in the study.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Manual Therapy Group: The treatment of this group consisted of two sessions per week, one hour each. We used joint traction, passive muscles stretching and Proprioceptive Neuromuscular Facilitation
  Manual Therapy: - 5 minutes. Termotherapy shalow to 50 cm away from the elbow, using a bulb of 250w.
  * 15 minutes. Joint traction of elbow, in submaximal mobility amplitude with distal fixation of humerus and proximal fixation of radius and ulna in neutral position of forearm. Joint traction in I-II degree of flexion and extension submaximal of elbow.
  * 15 minutes. Passive muscle stretching (within the limits of mobility). Compression technique, passive muscle stretching and relaxation in biceps and triceps.
  * 15 minutes. Proprioceptive neuromuscular facilitation (PNF) of upper limb.
  * 10 minutes. Local cryotherapy with ice bag and protection between it and the skin
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 9 | 9 | 9
degrees
  Pretreatment assessment | 138.31 (16.103) | 136.13 (14.818) | 138.00 (19.958)
  Postreatment assessment | 135.56 (16.66) | 140.31 (11.24) | 138.43 (18.47)
  Follow up assessment | 139.19 (16.64) | 140.31 (14.44) | 138.07 (17.39)

2. Primary Outcome: Changes in the Circumference of Arm
Description: Measurement of the arm circumference (in cm) at baseline as a result of hemophilic arthropathy and after treatment and follow-up. The measurement in the upper third of the arm, in the middle of the triceps muscle belly, with a tape measure. We use this outcome to measure circumference of the arm, it is the most clinical measurement used by physiotherapists.
Time Frame: as for outcome 1
Population: It has made an analysis by intention to treat with the 27 patients included in the study
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 9 | 9 | 9
cm
  Pretreatment assessment | 31.125 (3.144) | 31.331 (3.474) | 32.007 (3.837)
  Postreatment assessment | 31.23 (3.22) | 31.72 (3.20) | 31.85 (3.56)
  Follow up assessment | 31.02 (3.13) | 30.96 (2.70) | 31.68 (4.11)

3. Primary Outcome: Changes in Biceps Strength
Description: Measured by the breaking test for patients with haemophilia with a score from 0 to 5 (where 0 indicates normal strength and 5 is the absence of muscle contraction).
Time Frame: as for outcome 1
Population: It has made an analysis by intention to treat with the 27 patients included in the study
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 9 | 9 | 9
points
  Pretreatment assessment | 0.000 (0.000) | 0.094 (0.272) | 0.143 (0.363)
  Postreatment assessment | 0.03 (0.12) | 0.00 (0.00) | 0.07 (0.18)
  Follow up assessment | 0.06 (0.17) | 0.00 (0.00) | 0.07 (0.18)

4. Primary Outcome: Changes in the Pain Perception of Elbow
Description: Using the visual analogue scale, VAS (subjective rating scale with a score from 0 to 10, where 0 indicates no pain and 10 the maximum pain imaginable by the patient).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 8 | 8 | 7
points
  Pretreatment assessment | 0.156 (0.301) | 0.719 (0.752) | 0.143 (0.305)
  Postreatment assessment | 0.09 (0.20) | 0.34 (0.43) | 0.07 (0.67)
  Follow up assessment | 0.18 (0.35) | 0.12 (0.28) | 0.10 (0.28)

5. Primary Outcome: Assessment of Radiological Joint Deterioration
Description: Pettersson scale is an additive scale that assesses the radiological joint damage in patients with hemophilic arthropathy. It is scored as a range of 0-13 points (0: no joint damage; 13: maximum joint damage). This scale assesses: osteoporosis, widened epiphyseal, irregularity of the chondral surface, joint space narrowing, subchondral cyst formation, joint margins erosion, joint incongruence and joint deformity (angulation and displacement)
Time Frame: Screening visit (pretreatment assessment)
Population: It has made an analysis by intention to treat with the 27 patients included in the study. It has been estimated the radiological joint damage means (and standard deviation) for elbow joint.
Measure: Mean (Standard Deviation); unit: points
Groups:
- Manual Therapy Group: The treatment of this group consisted of two sessions per week, one hour each. We used joint traction, passive muscles stretching and Proprioceptive Neuromuscular Facilitation
  Manual Therapy: - 5 minutes. Termotherapy shalow to 50 cm away from the elbow, using a bulb of 250w.
  * 15 minutes. Joint traction of elbow. Joint traction in I-II degree of flexion and extension submaximal of elbow.
  * 15 minutes. Passive muscle stretching (within the limits of mobility). Compression technique, passive muscle stretching and relaxation in biceps and triceps.
  * 15 minutes. Proprioceptive neuromuscular facilitation (PNF) of upper limb, from the abduction, flexion and external rotation of shoulder with extension of elbow and dorsal flexion of wrist.
  * 10
Arm/Group | Manual Therapy Group | Educational Gruop | Control Group
Number analyzed (Participants) | 9 | 9 | 9
points | 9.63 (1.62) | 8.50 (3.40) | 7.57 (2.90)

6. Secondary Outcome: Characteristics of the Patients
Description: Age of patients included in teh study (years)
Time Frame: Screening visit (pretreatment assessment)
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 9 | 9 | 9
years | 33.78 (15.72) | 32.33 (11.67) | 37.33 (12.26)

7. Secondary Outcome: Frequency of Elbow Hemarthrosis
Description: Number of elbow hemarthrosis in the month prior to study
Time Frame: Screening visit (pretreatment assessment)
Measure: Mean (Standard Deviation); unit: bleeding events
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Number analyzed (Participants) | 9 | 9 | 9
bleeding events
  Hemarthros the month before the beginning of the s | 1.06 (1.23) | 1.06 (0.68) | 0.71 (0.91)
  Hemarthros during the study | 0.00 (0.00) | 0.00 (0.00) | 0.62 (0.87)

ADVERSE EVENTS:
Arm/Group | Educational Gruop | Manual Therapy Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
A limitation of our study is the low sample size (n = 27), although 96% of paients who met the inclusion criteria participated Due to the randomization of subjects there was no division proportionate according to the severity of haemophilia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No